CLINICAL TRIAL: NCT01688921
Title: Jet Injection for Influenza: A Randomized Controlled Clinical Trial to Demonstrate Non Inferiority of Jet Injection vs. Needle and Syringe for Administration of Trivalent Inactivated Influenza Vaccine
Brief Title: Jet Injection for Influenza
Acronym: JIFI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PharmaJet, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PJ-501-12-2
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-09

CONDITIONS: Influenza, Human
Keywords: Injections, Jet; Influenza Vaccines
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- STRATIS Needle-Free (Experimental): Patients assigned to this arm will receive AFLURIA vaccine administered using the Stratis needle-free injection device.
  Interventions: Biological: AFLURIA vaccine (2012-2013 formulation); Device: Needle-Syringe; Device: Stratis needle-free injection device
- Needle-Syringe (Active Comparator): Patients assigned to this arm will receive AFLURIA vaccine administered using a needle and syringe.
  Interventions: Biological: AFLURIA vaccine (2012-2013 formulation); Device: Needle-Syringe; Device: Stratis needle-free injection device

INTERVENTIONS:
Biological: AFLURIA vaccine (2012-2013 formulation) — Patients will receive a single 0.5 mL injection of AFLURIA vaccine in the deltoid region.
  Other Names: trivalent inactivated influenza vaccine (TIV); influenza virus vaccine
Device: Needle-Syringe
Device: Stratis needle-free injection device

SUMMARY:
The purpose of this study is to determine if the administration of a seasonal flu vaccine using a PharmaJet's needle-free injection device (STRATIS) is equivalent to needle and syringe administration, as measured by laboratory tests of immune response.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 and ≤64 years of age at the time of enrollment
* Willing and able to give informed consent after reading the consent form and adequate opportunity to discuss the study with the investigator or qualified designee
* Willing and able to adhere to all protocol required study procedures and to attend scheduled visits.
* Able to receive the TIV influenza vaccine, based on University of Colorado Health (UCH) employee health flu screening guidelines.
* Stable health status with no exclusionary medical or neuropsychiatric conditions as determined during the screening evaluation and based on the clinical judgment of the investigator or qualified designee.
* Access to a consistent means of telephone contact

Exclusion Criteria:

* Presence of any febrile illness (oral temperature >38°C) on the day of immunization. Such subjects will be reevaluated for enrollment after resolution of illness.
* Presence of significant acute or chronic uncontrolled medical or neuropsychiatric illness and /or presence of any significant condition that may prohibit inclusion as determined by the investigator or his qualified designee. Uncontrolled is defined as: requiring institution of a new treatment within 1 month prior to study enrollment or change in medication dosage in the month prior to study enrollment.
* Any immunosuppressive condition including: history of HIV infection, cancer or cancer treatment within 3 years of study enrollment, systemic glucocorticoids (in a dose ≥10 mg prednisone daily or equivalent for more than 7 consecutive days or for 10 or more days in total) within 1 month of study enrollment, or any other cytotoxic or immunosuppressive drug within 3 months of study enrollment. Any significant disorder of coagulation that would increase the risk of intramuscular injections or treatment with Coumadin derivatives or heparin.
* Known or suspected to be allergic to eggs, chicken protein, gentamicin or influenza vaccine.
* History of severe or previous serious adverse reaction after an influenza vaccination.
* Receipt of any immunoglobulin and/or blood products within 3 months of immunization or planned administration of any of these products during the study period.
* Prior history of any demyelinating disease including Guillain-Barre syndrome.
* Presence of an active neurological disorder.
* History of significant alcohol or drug abuse within one year prior to study enrollment.
* Influenza vaccination or laboratory confirmed influenza infection within the previous six months before study vaccination or planned influenza vaccination during the study period.
* Planned administration of any non-influenza vaccines 30 days prior to the study or during the study period.
* Pregnant or plans to become pregnant during the study period.
* Currently enrolled in another vaccine or drug study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1250 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David K Cobb, MD, MPH, Principal Investigator — Rocky Mountain Infectious Disease Consultants; Linda McAllister, MD, PhD, Study Director — PharmaJet, Inc.
Locations (3):
- United States (3):
  - Poudre Valley Hospital, Fort Collins, Colorado
  - University of Colorado Health Harmony Campus, Fort Collins, Colorado
  - Medical Center of the Rockies, Loveland, Colorado

REFERENCES:
- [Derived] McAllister L, Anderson J, Werth K, Cho I, Copeland K, Le Cam Bouveret N, Plant D, Mendelman PM, Cobb DK. Needle-free jet injection for administration of influenza vaccine: a randomised non-inferiority trial. Lancet. 2014 Aug 23;384(9944):674-81. doi: 10.1016/S0140-6736(14)60524-9. Epub 2014 May 31. PMID 24881803

RESULTS

PARTICIPANT FLOW:
Groups:
- STRATIS: Patients assigned to this arm will receive AFLURIA vaccine administered using the STRATIS needle-free injection device.
  AFLURIA vaccine (2012-2013 formulation): Patients will receive a single 0.5 mL injection of AFLURIA vaccine in the deltoid region.
  STRATIS needle-free injection device
- Needle-Syringe: Patients assigned to this arm will receive AFLURIA vaccine administered using a needle and syringe.
  AFLURIA vaccine (2012-2013 formulation): Patients will receive a single 0.5 mL injection of AFLURIA vaccine in the deltoid region.
  Needle-Syringe
Period: Overall Study
Arm/Group | STRATIS | Needle-Syringe
Started | 627 | 623
Completed | 611 | 608
Not Completed | 16 | 15
Not completed — Lost to Follow-up | 7 | 13
Not completed — Physician Decision | 6 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — informed consent | 3 | 0

BASELINE CHARACTERISTICS:
Population: Three subjects randomized to the PJ Stratis arm did not have properly documented informed consent and were excluded from the Full Analysis Set (FAS).
Groups:
- Total: Total of all reporting groups
Arm/Group | STRATIS | Needle-Syringe | Total
Number analyzed (Participants) | 624 | 623 | 1247
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.3 (12.92) | 41.5 (12.49) | 41.4 (12.70)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 624 | 623 | 1247
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 449 | 432 | 881
  Male | 175 | 191 | 366
Region of Enrollment [Number; unit: participants]
  United States | 624 | 623 | 1247

OUTCOME MEASURES:

1. Primary Outcome: Anti Influenza Type A/H1N1 Hemagglutination Inhibition (HAI) Antibody Geometric Mean Titer (GMT)
Description: The GMT criterion for non-inferiority for the upper limit of the 95% CIs of the GMT ratio(GMT with NS / GMT with PJ Stratis) for A/H1N1 antigen will not exceed 1.5 fold.
Time Frame: 28 days
Population: The immunogenicity analyses were conducted using data from subjects in the Immunogenicity Population.
Measure: Geometric Mean (Standard Deviation); unit: Titers
Groups:
- PJ STRATIS: Patients assigned to this arm will receive AFLURIA vaccine administered using the PJ STRATIS needle-free injection device.
  AFLURIA vaccine (2012-2013 formulation): Patients will receive a single 0.5 mL injection of AFLURIA vaccine in the deltoid region.
  PJ STRATIS needle-free injection device
Arm/Group | PJ STRATIS | Needle-Syringe
Number analyzed (Participants) | 562 | 568
Titers
  Day 0 | 4.43 (1.348) | 4.38 (1.352)
  Day 28 | 5.64 (1.006) | 5.64 (0.997)
Statistical Analysis 1: Comparison: PJ STRATIS vs Needle-Syringe; For a sample size of 550 per group each test has an individual power of > 99% to rule out the 1.5-fold difference using a two-sided α = 0.05, assuming equal GMTs between the two treatment groups. The overall power for the study to demonstrate the non-inferiority for the 6 co-primary endpoints is > 80%, computed as product of 6 individual powers; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was defined as the upper bound of the two-sided 95% CI of the GMT ratio (GMT with NS / GMT with PJ Stratis) for each antigen did not exceed 1.5 fold; Geometric Mean Ratio = 0.99, 95% CI 2-sided [0.88 to 1.12]

2. Primary Outcome: Anti Influenza Type A/H2N3 Hemagglutination Inhibition (HAI) Antibody Geometric Mean Titer (GMT)
Description: The GMT criterion for non-inferiority for the upper limit of the 95% CIs of the GMT ratio(GMT with NS / GMT with PJ Stratis) for each antigen to not exceed 1.5 fold.
Time Frame: 28 days
Population: The immunogenicity analyses were conducted using data from subjects in the Immunogenicity Population.
Measure: Geometric Mean (Standard Deviation); unit: Titers
Groups:
- PJ STRATIS: Patients assigned to this arm will receive AFLURIA vaccine administered using the STRATIS needle-free injection device.
  AFLURIA vaccine (2012-2013 formulation): Patients will receive a single 0.5 mL injection of AFLURIA vaccine in the deltoid region.
  PJ STRATIS needle-free injection device
Arm/Group | PJ STRATIS | Needle-Syringe
Number analyzed (Participants) | 562 | 568
Titers
  Day 0 | 4.22 (1.283) | 4.32 (1.290)
  Day 28 | 5.51 (1.022) | 5.58 (0.987)
Statistical Analysis 1: Comparison: PJ STRATIS vs Needle-Syringe; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 1.08, 95% CI 2-sided [0.96 to 1.21]

3. Primary Outcome: Anti Influenza Type B Hemagglutination Inhibition (HAI) Antibody Geometric Mean Titer (GMT)
Description: as for outcome 2
Time Frame: 28 days
Population: The immunogenicity analyses were conducted using data from subjects in the Immunogenicity Population.
Measure: Geometric Mean (Standard Deviation); unit: Titers
Arm/Group | PJ STRATIS | Needle-Syringe
Number analyzed (Participants) | 562 | 568
Titers
  Day 0 | 2.60 (1.028) | 2.54 (1.003)
  Day 28 | 3.75 (1.037) | 3.68 (1.061)
Statistical Analysis 1: Comparison: PJ STRATIS vs Needle-Syringe; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 0.94, 95% CI 2-sided [0.83 to 1.06]

4. Primary Outcome: Anti Influenza Type A/H1N1 Seroconversion
Description: Seroconversion is defined as a 4-fold rise in HAI titer in post-immunization serum relative to pre-immunization serum, or if pre-immunization serum had an undetectable titer (<1:10), attainment of a post-immunization titer of ≥1:40.
Time Frame: 28 days
Population: The immunogenicity analyses were conducted using data from subjects in the Immunogenicity Population.
Measure: Number; unit: Percent of Participants
Arm/Group | PJ STRATIS | Needle-Syringe
Number analyzed (Participants) | 562 | 568
Percent of Participants | 37.5 | 38.4
Statistical Analysis 1: Comparison: PJ STRATIS vs Needle-Syringe; For a sample size of 550 per group each test has an individual power of > 95% to rule out the 10 percentage points difference using a one-sided α = 0.025, assuming equal seroconversion rates between the two treatment groups. The overall power for the study to demonstrate the non-inferiority for the 6 co-primary endpoints is > 80%, computed as product of 6 individual powers; Test type: Non-Inferiority or Equivalence — Seroconversion rate defined as the proportion of subjects with either a pre-vaccination titer of <10 achieving a post-vaccination antibody of HI titer of ≥ 40 or with a pre-vaccination HI titer of ≥ 10 achieving a four-fold or greater increase in post-vaccination HI titer. The non-inferiority margin was defined as the upper bound of the two-sided 95% CI on the difference between the seroconversion rates (rate with NS - with PJ Stratis) for each vaccine strain did not exceed 10 percentage points; Seroconversion Rate Difference = 0.8, 95% CI 2-sided [-4.8 to 6.5]

5. Primary Outcome: Anti Influenza Type A/H3N2 Seroconversion
Description: as for outcome 4
Time Frame: 28 days
Measure: Number; unit: Percent of Participants
Arm/Group | PJ STRATIS | Needle-Syringe
Number analyzed (Participants) | 562 | 568
Percent of Participants | 43.8 | 45.1
Statistical Analysis 1: Comparison: PJ STRATIS vs Needle-Syringe; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — Seroconversion rate defined as the proportion of subjects with either a pre-vaccination titer of <10 achieving a post-vaccination antibody of HI titer of ≥ 40 or with a pre-vaccination HI titer of ≥ 10 achieving a four-fold or greater increase in post-vaccination HI titer. The non-inferiority margin was defined as the upper bound of the two-sided 95% CI on the difference between the seroconversion rates(rate with NS - with PJ Stratis) for each vaccine strain did not exceed 10 percentage points; Seroconversion Rate Difference = 1.3, 95% CI 2-sided [-4.5 to 7.1]

6. Primary Outcome: Anti Influenza Type B Seroconversion
Description: as for outcome 4
Time Frame: 28 days
Population: The immunogenicity analyses were conducted using data from subjects in the Immunogenicity Population.
Measure: Number; unit: Percent of Participants
Arm/Group | PJ STRATIS | Needle-Syringe
Number analyzed (Participants) | 562 | 568
Percent of Participants | 34.9 | 35.2
Statistical Analysis 1: Comparison: PJ STRATIS vs Needle-Syringe; For a sample size of 550 per group each test has an individual power of > 91% to rule out the 10 percentage points difference using a one-sided α = 0.025, assuming equal seroconversion rates between the two treatment groups. The overall power for the study to demonstrate the non-inferiority for the 6 co-primary endpoints is > 80%, computed as product of 6 individual powers; Test type: Non-Inferiority or Equivalence — Seroconversion rate was defined as the proportion of subjects with either a pre-vaccination titer of <10 achieving a post-vaccination antibody of HI titer of ≥ 40 or with a pre-vaccination HI titer of ≥ 10 achieving a four-fold or greater increase in post-vaccination HI titer. The upper-bound of the two-sided 95% CI on the difference in seroconversion rates for the A/H1N1, A/H3N2, and B strains did not exceed 10 percentage points (6.5, 7.1, and 5.9 respectively); Seroconversion Rate Difference = 0.3, 95% CI 2-sided [-5.2 to 5.9]

7. Secondary Outcome: Number of Subjects With Complaints Within 30 Minutes Following Vaccination
Time Frame: Within 30 minutes post-vaccination
Population: The safety population included 1247 subjects (N=624 PJ Stratis, N=623 NS).
Measure: Number; unit: participants
Arm/Group | PJ STRATIS | Needle-Syringe
Number analyzed (Participants) | 624 | 623
participants
  Pain | 163 | 69
  Tenderness | 104 | 36
  Itching | 63 | 17
  Redness | 113 | 11
  Swelling | 5 | 0
  Bruising | 0 | 0
Statistical Analysis 1: Comparison: PJ STRATIS vs Needle-Syringe; Test type: Non-Inferiority or Equivalence — Immediate adverse events were reported within 30 minutes of receiving the vaccination; therefore, they are all considered related to study treatment; p < 0.001, Fisher Exact

8. Secondary Outcome: Number of Subjects With Vaccine Reactogenicity Events
Description: Vaccine reactogenicity will be collected on a patient-completed diary card during checkout from Day 0 and on the next six evenings post-vaccination. The following adverse events will be solicited on the diary card: pain at injection site, tenderness at injection site, redness where the injection is given; induration/swelling (lump) where the injection is given; bruising where the injection is given; itching where the injection is given; headache; tiredness/fatigue (asthenia, lethargy, malaise); general muscle ache (myalgia); chills; nausea; vomiting. Subjects will also record their oral temperature on the diary card each evening.
Time Frame: Day 0, 1, 2, 3, 4, 5, and 6
Population: The safety population included 1247 subjects (N=624 PJ Stratis, N=623 NS). Eight subjects (624-616) in the PJ Stratis group and 16 (623-607) in the NS group did not return the 7-Day Diary Card.
Measure: Number; unit: participants
Arm/Group | PJ STRATIS | Needle-Syringe
Number analyzed (Participants) | 616 | 607
participants
  Pain | 397 | 299
  Tenderness | 551 | 472
  Itching | 151 | 50
  Redness | 366 | 115
  Swelling | 392 | 115
  Bruising | 107 | 32
  Headache | 151 | 133
  Malaise | 191 | 171
  Myalgia | 222 | 214
  Chills | 43 | 43
  Nausea | 40 | 39
  Vomiting | 8 | 11
Statistical Analysis 1: Comparison: PJ STRATIS vs Needle-Syringe; Test type: Non-Inferiority or Equivalence — The safety population included subjects who received the vaccination and for whom follow-up data were available for a specific safety analysis. Therefore, the denominators for different safety tables vary, depending on the availability of the data; p < 0.001, Fisher Exact

9. Secondary Outcome: Number of Subjects With Spontaneously Reported Adverse Events
Description: Subjects will be asked to report any other symptoms experienced in addition to the solicited "immediate" and "vaccine reactogenicity" events. Any other events reported will be tabulated as spontaneously reported adverse events.
Time Frame: 28 days
Population: The safety population included 1247 subjects (N=624 PJ Stratis, N=623 NS).
Measure: Number; unit: participants with spontaneous AEs
Arm/Group | PJ STRATIS | Needle-Syringe
Number analyzed (Participants) | 624 | 623
participants with spontaneous AEs | 92 | 73

10. Secondary Outcome: Percentage of Subjects Who Received a PJ Stratis Injection Would Choose to Receive This Type of Injection Again
Time Frame: 28 Days
Population: Safety population
Measure: Number; unit: Percent of Participants
Arm/Group | PJ STRATIS
Number analyzed (Participants) | 624
Percent of Participants | 89

ADVERSE EVENTS:
Time Frame: Immediate complaints were solicited from subjects in the safety population following vaccination: pain, tenderness, itching, redness, swelling, and bruising at the vaccination site.
Description: Solicited adverse events were those events specifically sought for and recorded by the subject in the 7-Day Diary Card.
  The denominators were determined for each individual AE for each summary window (Day 0-3 or 4-6). Subjects in Safety Populations were excluded from the denominator if there was no data captured for the AE within summary window.
Arm/Group | STRATIS | Needle-Syringe
Serious Adverse Events (participants affected / at risk) | 1/624 | 2/623
Other Adverse Events (participants affected / at risk) | 586/624 | 516/623
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STRATIS (N=624) | Needle-Syringe (N=623)
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 1 | 0 — The SAE was unrelated to subject's participation in the study.
Peritonitis (Infections and infestations) | 1 | 0 — The SAE reported was unrelated to subject's participation in the study.
Viral Meningitis (Infections and infestations) | 0 | 1 — The SAE reported was unrelated to the subject's participation in the study.
Coronary Artery Disease (Cardiac disorders) | 0 | 1 — The SAE reported was unrelated to the subject's participation in the study.
Myocardial Infarction (Cardiac disorders) | 0 | 1 — The SAE reported was unrelated to the subject's participation in the study.
Arterial Injury (Cardiac disorders) | 0 | 1 — The SAE reported was unrelated to the subject's participation in the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | STRATIS (N=624) | Needle-Syringe (N=623)
Pain (General disorders) | 397/616 | 299/606 — Local symptoms at injection site within 6 days of vaccination with Grade of >=1
Tenderness (General disorders) | 551/616 | 471/606 — Local Adverse Reaction within 6 days of vaccination and Grade of >=1
Itching (General disorders) | 146/540 | 49/527 — Local Adverse Reaction occurring within 6 days of vaccination and a Grade of >=1
Redness (General disorders) | 366/609 | 115/599 — Local event occurring within 6 days of vaccination and Grade of >=1
Swelling (General disorders) | 392/605 | 118/599 — Local Adverse Reaction occurring within 6 days of vaccination with Grade level >=1
Bruising (General disorders) | 104/607 | 30/599 — Local Adverse Reaction occurring within 6 days of vaccination with Grade level of >=1
Myalgia (Musculoskeletal and connective tissue disorders) | 222/610 | 214/602
Headache (Nervous system disorders) | 151/612 | 133/603
Malaise (Immune system disorders) | 191/612 | 171/602
Chills (Nervous system disorders) | 43/610 | 43/601
Nausea (Gastrointestinal disorders) | 40/610 | 39/601

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less